CLINICAL TRIAL: NCT05075447
Title: Diagnosis and Treatment Plan for Destructive and Conduct Disorder Children With Indifferent Traits and Emotion Regulation
Brief Title: Treatment Plan for ADHD With Indifferent Traits
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XH-21-007
Record Dates: First submitted 2021-07-23; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-03

CONDITIONS: Lack of; Attention, With Hyperactivity (ADHD)
Keywords: Destructive; CD; Apathy; Emotion regulation; Treatment
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Lethargy; Emotional Regulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ADHD group (Experimental): Child diagnosed with ADHD
  Interventions: Behavioral: Emotion Control Treatment Program
- control group (No Intervention): Children without any diagnosis
- ADHD+ODD/CD group (Experimental): Child diagnosed with ADHD+ODD/CD
  Interventions: Behavioral: Emotion Control Treatment Program

INTERVENTIONS:
Behavioral: Emotion Control Treatment Program — Intervention programs include Child Training and Training in real scenes
  Arms: ADHD group; ADHD+ODD/CD group

SUMMARY:
For children with ADHD aged 4-10 at the time of enrollment, starting from preschool, focusing on apathy and emotional control, using psycho-behavioral measurements, EEG experiments, and eye tracking technology to evaluate and implement targeted Sexual intervention and six-month follow-up. Establish a diagnosis and treatment decision analysis model and psychological treatment plan for ODD/CD.

DETAILED DESCRIPTION:
Destructive, conduct disorder children have emotional processing defects, including apathy and ruthless traits, emotional disorders, may be early diagnosis of conduct disorder (Conduct Disorder, CD) or attention deficit hyperactivity disorder (Attention Deficit Hyperactivity Disorders, ADHD) comorbid CD sensitivity Sexual indicators, systemic psychotherapy for these children's indifference characteristics and emotional disorders will improve related symptoms. This study will start with preschool children with ADHD, design evaluation indicators for emotional traits for children aged 4-10, combined with various psychological evaluations, and use advanced brain electricity combined with eye tracking research technology to provide candidate indicators for evaluation; and On the basis of previous research, establish a treatment plan to improve pathological emotional characteristics and emotional disorders; establish a predictive intervention decision model from preschool to school-age ADHD comorbid CD to provide methods for precise diagnosis and treatment options. The early prevention and intervention of ADHD and CD has practical significance and maneuverability.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 years, 0 months and 10 years old and 11 months old, who have been diagnosed by a doctor who is at least the attending physician in the pediatric psychiatric department and meet the American Diagnostic and Statistical Manual of Mental Disorders (Fifth Edition) ADHD diagnostic criteria, have a total IQ higher than 80, and the subjects are doing this The baseline level of the study has not received any medical treatment before.

Exclusion Criteria:

* Attention deficit disorder caused by organic diseases of the nervous system, extensive developmental disorders, mental retardation, childhood schizophrenia, mood disorders, epilepsy, and other organic diseases or other primary mental disorders; exclude parents or guardians from suffering Severe mental illness, such as schizophrenia, mood disorders (onset period), etc., and a degree below junior high school.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Apathy and ruthlessness（CU traits） of 60 children with ADHD | Collected when the case is enrolled
  The CU traits of children with ADHD assessed by A CU questionnaire tests.
Apathy and ruthlessness（CU traits） of 60 children with ADHD+ODD/CD | Collected when the case is enrolled
  The CU traits of children with ADHD assessed by A CU questionnaire tests.

SECONDARY OUTCOMES:
The executive function in real life of 120 children with ADHD | through the intervention completion, an average of 8 weeks
  The executive function in real life of 120 children with ADHD assessed by BRIEF

CONTACTS AND LOCATIONS:
Overall Officials: Jingyi Wu, Master, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai, China